CLINICAL TRIAL: NCT05122858
Title: EUS-guided Biliary Drainage of First Intent With the Lumen Apposing Metal Stent vs. ERCP in the Management of Malignant Distal Biliary Obstruction: a Randomized Controlled Trial.
Brief Title: EUS-guided Biliary Drainage of First Intent With the Lumen Apposing Metal Stent vs. ERCP in the Management of Malignant Distal Biliary Obstruction (AXIOS-CPRE)
Acronym: AXIOS-CPRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A00654-35
Record Dates: First submitted 2021-11-04; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography; Biliary Drainage; Echography Ultrasound
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS guided biliary drainage (Experimental)
  Interventions: Procedure: EUS guided biliary drainage
- ERCP (Endoscopic Retrograde Cholangiopancreatography (Active Comparator)
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: EUS guided biliary drainage — A curvilinear endoscope is inserted orally and advanced to the duodenal bulb. Biliary accessibility will then be confirmed via endoscopic ultrasound (EE) from the duodenal bulb and via Doppler ultrasound to exclude any disturbing vessels. In order to maintain the stability of the duodenal bulb, the long endoscope position will be used whenever possible. A SMAL (AxiosTM) will be inserted with the assistance of cautery and then deployed. The use of a guidewire and the choice of stent size will be at the endoscopist's discretion.
  Arms: EUS guided biliary drainage
Procedure: ERCP — A duodenoscope is advanced to the papilla orally. The bile duct is then cannulated with a sphincterotome using the guidewire assisted technique. A cholangiogram is then performed followed by the placement of a self-expanding metallic bile stent. The performance of the biliary sphincterotomy before placement of the stent and the choice of the size of the stent will be at the discretion of the endoscopist.
  Arms: ERCP (Endoscopic Retrograde Cholangiopancreatography

SUMMARY:
The main objective is to compare the EUS-BD with the insertion of a LAMS vs. traditional ERCP to restore biliary patency. Although ERCP has been the primary treatment for many years, it is associated with a significant risk of procedural complications and possible stent blockage. EUS-BD has been shown to be potentially safer and is associated with a lower risk of stent blockage. We seek with our study to determine whether EUS-BD may be the most effective treatment modality.

ELIGIBILITY:
Inclusion Criteria:

* Radiological diagnosis (with or without pathological diagnosis) of a malignant obstruction of the borderline resectable distal bile ducts, locally advanced or unresectable distal to the hilum, at a minimum distance of 2 cm.
* Resectability based on tumor staging after axial imaging and evaluation by a physician (surgeon, oncologist and / or gastroenterologist).
* High results of the liver function test with a serum bilirubin level at least 3 times above the upper limit of normal (18.9 μmol / L)
* Dilated extrahepatic bile duct measuring at least 1.2 cm in axial imaging, ultrasound or endoscopy.
* Karnofsky index> 30%
* ASA score <IV
* Patient accepting the constraints of research
* Patient affiliated or beneficiary of a social security scheme
* Patient having signed an informed consent

Exclusion Criteria:

* - Hilar obstruction (biliary obstruction located <2 cm from the hilum)
* Coagulopathy and / or thrombocytopenia that cannot be corrected
* Age <18 years old
* Liver metastases involving> 30% of hepatic volume
* Liver cirrhosis with portal hypertension or ascites
* Biliary sphincterotomy or placement of a stent performed in the past
* Anatomy modified by surgery
* Common bile ducts measuring less than 1.2 cm will be excluded.
* Patient with clinical and radiological signs of stenosis of the gastric outlet
* Patient participating in another clinical study
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant, breastfeeding or parturient woman
* Patient hospitalized without consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Number of participant with stent dysfunction (obstruction or migration) requiring endoscopic, radiological or surgical intervention | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé des Peupliers, Paris, France